CLINICAL TRIAL: NCT01510990
Title: First Line Gefitinib Treatment for Advanced Non-small Cell Lung Cancer (NSCLC) by the FDG-PET Metabolic Response
Brief Title: First Line Gefitinib by FDG-PET Metabolic Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sang-We Kim, Principal Investigator, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2011-0858
Record Dates: First submitted 2012-01-10; First posted 2012-01-18 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Gefitinib; FDG-PET
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib (Experimental): After a baseline 18F FDG-PET, patients are treated with gefitinib 250mg/d as 1st line treatment for 7 days. And follow up 18F-FDG PET image is acquired after 1 week's treatment of gefitinib (with window period +/- 2 days).
  If % decrease of peak SUV of main lesion is 20% or more, gefitinib treatment is continued till progression, unacceptable toxicities or patient's refusal. But if % decrease of peak SUV of main lesion less than 20% or peak SUV increase, gefitinib treatment is stopped, and changed to Pemetrexed/Cisplatin chemotherapy.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — gefitinib 250mg/day daily
  Other Names: Iressa

SUMMARY:
When considering 1st line gefitinib treatment for NSCLC, the investigators need epidermal growth factor receptor (EGFR) mutational status of the tumor. But most patients do not give us such information at the time of diagnosis, because it requires tumor tissue and some time period for EGFR examination. So, investigators develop a protocol of 1st line gefitinib treatment for NSCLC according to FDG-PET response. If a patient shows 20% or more decrease of peak standard uptake value (SUV) after 1 week's gefitinib treatment, he or she will be continued the treatment. If a patient shows less than 20% decrease of SUV, he or she will be switched to other chemotherapy.

DETAILED DESCRIPTION:
Gefitinib has anti-tumor activity as a result of EGFR tyrosine kinase inhibition, reducing multiple downstream signaling processes that activate cell proliferation and other cell responses, including cell migration angiogenesis, and reduced apoptosis. Recently, it has been approved for the first line treatment of advanced NSCLC that harbors EGFR mutation. In IPASS trial, tumors with EGFR mutation produced 71.2% of clinical response to first line gefitinib while tumors with wild type EGFR showed only 1.1% of response. Therefore, patient selection is critical for the clinical use of EGFR tyrosine kinase inhibitors as first line treatment.

When considering 1st line gefitinib treatment for NSCLC, we need EGFR mutational status of the tumor. But most patients do not give us such information at the time of diagnosis, because it requires tumor tissue and some time period for EGFR examination. So, we need other strategies such as using PET scan for early prediction of response to gefitinib.

Glucose metabolic activity closely reflects responses to gefitinib therapy. In preclinical study with gefitinib sensitive cell lines, there was a dramatic decrease in FDG uptake as early as 2 hours after treatment. And these metabolic alterations preceded changes in cell cycle distribution, thymidine uptake and apoptosis. In contrast, gefitinib resistant cells exhibited no measurable changes in FDG uptake, either in cell culture or in vivo.

The strategy using FDG-PET may guide us to perform 1st line geftinib. Recently investigators reported that FLT-PET or FDG-PET could predict response to EGFR tyrosine kinase (TKI) early after 1 week of treatment. And % decrease more than 20% of maximum SUV of main lesion after 1 week of EGFR TKI treatment could predict response to that drug. More than 20% decrease of SUV is a significant change during reproducibility test and also considered as a criteria for response prediction of paclitaxel/cisplatin chemotherapy.

So, investigators develop a protocol of 1st line gefitinib treatment for NSCLC according to FDG-PET response. And if the patient showed less than 20% decrease of peak SUV, investigators will stop gefitinib and treat him or her with the regimen of pemetrexed/cisplatin.

ELIGIBILITY:
Inclusion criteria

* More than 18 years of age
* Advanced or metastatic adenocarcinoma of the lung. Non-smoking or light smoking patients (less than 10 PY smoking and more than 10 years of ex-smoking period) are preferred to enrich the patients with clinical response to gefitinib.
* Chemonaive patients.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or and which is suitable for accurate repeated measurements.
* ECOG PS 0-2
* Patients with tissue for the detection of EGFR mutation
* At least 1 week since the last radiotherapy. Patients must have recovered from all acute toxicities from radiotherapy.
* Patients must have adequate hematologic, renal and liver function as defined by Hb > 9g/dL, neutrophils > 1000/mm3, platelets > 50,000/mm3, creatinine < 2mg/dL, and AST (SGOT) and/or ALT (SGPT) < 5 x UNL (upper normal limit).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Written and voluntary informed consent understood, signed and dated.

Exclusion criteria

* Symptomatic brain metastasis. Brain metastases stable < 2 weeks before dosing or requiring concurrent steroid treatment or with clinical symptoms.
* Major surgery within 3 weeks prior to study enrollment.
* Previous (less than 3 years ago) or current malignancies at sites other than curatively treated in situ carcinoma of cervix, or basal or squamous cell carcinoma of the skin.
* Past medical history of interstitial lung diseas, drug induced interstitial disease, radiation pneumonitis which required steroid treatment or any active interstitial lung disease.
* Pre-existing idiopathic pulmonary fibrosis on CT scans on baseline.
* Insufficient lung function as determined by either clinical examination or an arterial oxygen tension (PaO2) < 70mmHg.
* Uncontrolled diabetes mellitus and FBS > 150mg/dL.
* Severe medical illness or active infection that would impair the ability to receive gefitinib.
* Pregnancy or breast feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate | one year
  The primary objective is to see the response rate of gefitinib in the patients who showed % decrease of peak SUV of main lesion 20% or more and continuously treated with gefitinib.

SECONDARY OUTCOMES:
Objective response rate by EGFR mutational status | One year
  The secondary object is to see the relationship of changes in FDG uptake after gefitinib treatment with EGFR mutation; sensitivity, specificity, positive predictive value, and negative predictive value will be calculated comparing the groupings created by FDG-PET and actual EGFR mutational status.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-We Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea